CLINICAL TRIAL: NCT02076802
Title: Regular Physical Exercise and Salt Diet Effect on Progression of Coronary Disease in Patients With Prehypertension
Brief Title: Regular Physical Exercise and Salt Diet on Coronary Artery Disease in Patients With Prehypertension(RESTRAIN Pre-HT)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, xin Zhao, professor, General Hospital of Shenyang Military Region
Other Study IDs: GHSY-20130814
Record Dates: First submitted 2014-02-25; First posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-02

CONDITIONS: Coronary Atherosclerosis; Cardiovascular Disease
Keywords: prehypertension; coronary atherosclerosis; cardiovascular disease
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases; Prehypertension | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- lifestyle counseling: physical exercises
  Interventions: Behavioral: physical exercises

INTERVENTIONS:
Behavioral: physical exercises

SUMMARY:
The epidemic data shows that prehypertension is associated with cardiovascular disease, and heavy dietary salt intake could improve the developing of hypertension. We detected the risk factors of coronary atherosclerosis of prehypertensive patients with different levels of salt intake.

The aim of this multicenter prospective, randomized controlled study is to evaluate regular physical exercise and salt diet effects on progression of coronary artery disease in patients with prehypertension.

ELIGIBILITY:
Inclusion Criteria:

aged 45-75 Admission systolic BP between 120 and 139mmHg or diastolic BP between 80 and 89mmHg coronary artery stenosis was 30%-70% -

Exclusion Criteria:

with a history of myocardial infarction, coronary revascularization, congenital heart disease and cerebrovascular diseases

-

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coronary atherosclerosis patients with prehypertension
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-07 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
fatal and nonfatal myocardial infarction, or coronary revascularization | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Shenyang Militaly Region, Shenyang, Liaoning, China